CLINICAL TRIAL: NCT00819169
Title: A Phase 1b/2 Open Label, Dose Escalation Study of AMG 655 in Combination With AMG 479 in Subjects With Advanced, Refractory Solid Tumors
Brief Title: QUILT-3.026: AMG 655 in Combination With AMG 479 in Advanced, Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision - subjects rolled over to protocol 20101116
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070411; QUILT-3.026 (Other: NantCell, Inc.)
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Locally Advanced; Metastatic Cancer; Non-Small Cell Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Sarcoma; Solid Tumors
Keywords: AMG 655; AMG 479; Apoptosis; Monoclonal Antibody; Tumor Necrosis Factor; Insulin-like Growth Factor
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Pancreatic Neoplasms; Sarcoma | interventions — ganitumab; conatumumab

ARMS (4):
- Part 1 Cohort 3 (Experimental): AMG 479 18 mg/kg IV plus AMG 655 15 mg/kg IV (day 1 of each Q3W cycle)
  Interventions: Biological: AMG 479; Biological: AMG 655
- Part 1 Cohort 1 (Experimental): AMG 479 18 mg/kg IV plus AMG 655 1 mg/kg IV (day 1 of each Q3W cycle)
  Interventions: Biological: AMG 479; Biological: AMG 655
- Part 1 Cohort 2 (Experimental): AMG 479 18 mg/kg IV plus AMG 655 3 mg/kg IV (day 1 of each Q3W cycle)
  Interventions: Biological: AMG 479; Biological: AMG 655
- Part 2 (Experimental): AMG 479 18 mg/kg IV plus AMG 655 15 mg/kg Q3W, or the MTD, as determined in Part 1 of the study
  Interventions: Biological: AMG 479; Biological: AMG 655

INTERVENTIONS:
Biological: AMG 479 — AMG 479 is an investigational, fully human, monoclonal antibody that binds with Insulin-like growth factor receptor type 1.
Biological: AMG 655 — AMG 655 is an investigational, fully human, monoclonal antibody that binds with TNF-related apoptosis-inducing ligand, DR 5.
  Other Names: AMG 655 is also known as conatumumab.

SUMMARY:
This is a multi-center, 2-part phase 1b/2 study of AMG 655 in combination with AMG 479 to be conducted in the United States and Spain.

Part 1 is a dose escalation segment to identify a dose of AMG 655 in combination with AMG 479 that is safe and tolerable.

Part 2 will evaluate the safety and estimate the efficacy of AMG 655 at the dose selected in Part 1 in combination with AMG 479 for the treatment of patients with advanced NSCLC (non-squamous histology; squamous histology), CRC, pancreatic cancer, ovarian cancer, and sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Histologically or cytologically confirmed, locally advanced or metastatic, treatment-refractory solid tumors
* Part 2: Histologically or cytologically confirmed, locally advanced or metastatic: NSCLC (squamous or non-squamous cell carcinoma; up to 2 prior treatment regimens), Colorectal Cancer (up to 2 prior treatment regimens), Pancreatic Cancer (up to 1 prior treatment regimen), Ovarian cancer (up to 2 prior treatment regimens), or Sarcoma (up to 2 prior treatment regimens), according to cohort availability
* Eastern Cooperative Group (ECOG performance status of 0 or 1
* Women or men ≥16 years of age
* Adequate hematology, renal, hepatic, coagulation and glycemic function.

Exclusion Criteria:

* Presence of uncontrolled central nervous system (CNS) disease
* Systemic chemotherapy, hormonal therapy, immunotherapy, experimental or approved anticancer proteins/antibodies therapy ≤28 days before enrollment.
* Prior treatment with death receptor agonists (including but not limited to rhApo2L/TRAIL [AMG951], apomab, mapatumumab, lexatumumab, CS-1008)
* Prior treatment with IGF receptor antagonists (including but not limited to CP-751, 871, MK0646, AVE1642 or IMC-A12)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-01-16 (Actual); Primary Completion 2011-08-10 (Actual); Study Completion 2011-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Chawla S, Tabernero, J, Kindler, H., Reckamp, K., Chiorean, E., Azad, N., Lockhard, A., Hsu, CP., Baker, N., Galimi, F., Beltran, P., Baselga, J..Anticancer activity of the type I insulin-like growth factor receptor antagonist, ganitumab, in combination with the death receptor 5 agonist, conatumumab.Targeted Oncology;Tabernero J, Chawla SP, Kindler H, Reckamp K, Chiorean EG, Azad NS, Lockhart AC, Hsu CP, Baker NF, Galimi F, Beltran P, Baselga J. Anticancer activity of the type I insulin-like growth factor receptor antagonist, ganitumab, in combination with the death receptor 5 agonist, conatumumab. Target Oncol. 2014 May 11. [Epub ahead of print]
- [Derived] Tabernero J, Chawla SP, Kindler H, Reckamp K, Chiorean EG, Azad NS, Lockhart AC, Hsu CP, Baker NF, Galimi F, Beltran P, Baselga J. Anticancer activity of the type I insulin-like growth factor receptor antagonist, ganitumab, in combination with the death receptor 5 agonist, conatumumab. Target Oncol. 2015 Mar;10(1):65-76. doi: 10.1007/s11523-014-0315-z. Epub 2014 May 11. PMID 24816908
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4317391/

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2 Cohort 1: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Non-squamous NSCLC
- Part 2 Cohort 2: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Squamous Non -Small Cell Lung Cancer (NSCLC)
- Part 2 Cohort 3: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Colorectal Cancer (CRC)
- Part 2 Cohort 4: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Pancreatic Cancer
- Part 2 Cohort 5: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Ovarian Cancer
- Part 2 Cohort 6: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Sarcoma
Period: Overall Study
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Started | 3 | 3 | 3 | 15 | 8 | 16 | 16 | 9 | 16
Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3
Not Completed | 3 | 3 | 3 | 12 | 8 | 16 | 16 | 9 | 13
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 1 | 1 | 5 | 1 | 4
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1 | 0 | 6 | 2 | 2 | 1
Not completed — Death | 1 | 1 | 3 | 8 | 5 | 7 | 9 | 4 | 7
Not completed — Ineligibility determined | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative Decision | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 2 Cohort 2: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) Squamous NSCLC
- Part 2 Cohort 3: AMG 479 18 mg/kg (Q3W) with AMG 655 15 mg/kg (Q3W) CRC
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 15 | 8 | 16 | 16 | 9 | 16 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part 1 and Part 2 were analyzed separately.
  years
    Part 1: number analyzed (Participants) | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 9
    Part 1 | 48.0 (20.9) | 65.3 (1.2) | 46.0 (4.4) |  |  |  |  |  |  | 53.1 (14.1)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 15 | 8 | 16 | 16 | 9 | 16 | 80
    Part 2 |  |  |  | 61.0 (10.3) | 67.0 (7.3) | 59.1 (11.0) | 60.2 (8.8) | 58.0 (15.8) | 51.3 (9.8) | 58.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For part 2 the full analysis population was used which included only those subjects that received investigational product.
  Participants
    number analyzed (Participants) | 3 | 3 | 3 | 15 | 7 | 16 | 16 | 9 | 15 | 87
    Female | 2 | 1 | 2 | 8 | 2 | 5 | 5 | 9 | 10 | 44
    Male | 1 | 2 | 1 | 7 | 5 | 11 | 11 | 0 | 5 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: For part 2 the full analysis population was used which included only those subjects that received investigational product.
  Participants
    number analyzed (Participants) | 3 | 3 | 3 | 15 | 7 | 16 | 16 | 9 | 15 | 87
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 6
    White | 2 | 3 | 3 | 12 | 5 | 13 | 13 | 8 | 14 | 73
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: Incidence of adverse events and clinical laboratory abnormalities defined as DLTs. Dose-limiting toxicities included any grade 3 or higher hematologic or nonhematologic toxicity related to conatumumab or the combination of conatumumab with ganitumab except for lymphocytopenia and anemia.
Time Frame: Time from first dose up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) is defined as confirmed complete response or partial response using modified Response Evaluation Criteria in Solid Tumors [RECIST]: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Time from first dose up to 24 months
Population: A subject was included in the analysis if they received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 15 | 7 | 16 | 16 | 9 | 15
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival is defined as the number of days from study day 1 (first dose of investigational product) to the first observation of disease progression (by modified RECIST; or clinical progression, whichever came first) or death due to any cause. Disease progression by RECIST is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: Time from first dose up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 15 | 8 | 16 | 16 | 9 | 16
months | 1.4 [1.1 to 15.4] | 4.9 [1.6 to 5.5] | 1.3 [1.1 to 2.4] | 1.6 [1.3 to 3.7] | 3.3 [1.9 to 5.4] | 1.5 [1.3 to 2.6] | 1.4 [1.2 to 2.3] | 2.8 [1.6 to 3.9] | 1.3 [1.2 to 1.7]

4. Secondary Outcome: To Evaluate Anti-AMG 655 Antibody Formation and Anti-AMG 479 Antibody Formation
Time Frame: Time from first dose up to 24 months
Population: Antibody Population = All subjects in the full analysis set tested for antibodies during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 1 | 2 | 1 | 11 | 5 | 13 | 7 | 7 | 10
Participants
  AMG 655 - Binding antibody positive at any time | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AMG 655 - Neutralizing antibody positive at any time | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AMG 479 - Binding antibody positive at any time | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  AMG 479 - Neutralizing antibody positive at any time | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: To Evaluate the Concentration Level of AMG 655
Description: Median, minimum, and maximum concentration of AMG 655 at specified time points.
Time Frame: Cycle 1 Day 1 end of infusion; Cycle 3 Day 1 end of infusion (each cycle is 28 days, each infusion is up to 1 hour)
Population: PK population = All subjects in the full analysis set who underwent blood sampling for PK evaluation during the study.
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 3 | 2 | 2 | 13 | 7 | 14 | 14 | 7 | 13
μg/mL
  Cycle 1-End of Infusion: number analyzed (Participants) | 3 | 1 | 2 | 2 | 1 | 10 | 11 | 4 | 13
  Cycle 1-End of Infusion | 17.5 [17.3 to 19.4] | 59.0 [59.0 to 59.0] | 313 [261 to 365] | 244 [240 to 247] | 266 [266 to 266] | 240 [115 to 319] | 224 [130 to 293] | 327 [275 to 341] | 247 [91.3 to 392]
  Cycle 3-End of infusion: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 4 | 1 | 2 | 4
  Cycle 3-End of infusion | 23.6 [23.6 to 23.6] | 62.3 [62.3 to 62.3] | 302 [302 to 302] | 448 [448 to 448] |  | 311 [233 to 380] | 253 [253 to 253] | 423 [356 to 490] | 371 [328 to 466]

6. Secondary Outcome: To Evaluate the Concentration Level of AMG 479
Description: Median, minimum, and maximum concentration of AMG 479 at specified time points.
Time Frame: Cycle 1 Day 1 end of infusion; Cycle 3 Day 1 end of infusion (each cycle is 28 days, each infusion is up to 1 hour)
Population: PK population = All subjects in the full analysis set who underwent blood sampling for PK evaluation during the study.
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 3 | 2 | 2 | 13 | 7 | 14 | 14 | 9 | 13
μg/mL
  Cycle 1-End of infusion: number analyzed (Participants) | 3 | 1 | 2 | 2 | 1 | 8 | 12 | 5 | 13
  Cycle 1-End of infusion | 272 [198 to 279] | 268 [268 to 268] | 303 [257 to 349] | 215 [193 to 237] | 297 [297 to 297] | 227 [130 to 634] | 236 [121 to 391] | 324 [248 to 439] | 254 [169 to 445]
  Cycle 3-End of Infusion: number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 3 | 4
  Cycle 3-End of Infusion | 308 [308 to 308] |  | 338 [338 to 338] | 404 [404 to 404] |  | 262 [205 to 364] | 249 [249 to 249] | 323 [300 to 381] | 365 [244 to 420]

7. Secondary Outcome: Time to Response
Description: Time to response is the time from study day 1 to the first observation of an objective response. Subjects without an objective response are excluded from the analysis of this endpoint. Objective response is defined as a tumor response assessment of either complete response or partial response per modified Response Evaluation Criteria in Solid Tumors (RECIST) and will be determined based on the Investigator-reported assessment only for subjects with measurable disease at baseline. Per RECIST v 1.1: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Time from first dose up to 24 months
Population: Because no subjects in Part 2, and only one subject in Part 1, had an objective response the analyses of time to response was not calculated.
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the number of days between the date of first objective response to the time of the first progressive disease (per modified Response Evaluation Criteria in Solid Tumors [RECIST] or clinical progression, whichever occurs first) or death due to any cause. Objective response is defined as a tumor response assessment of either complete response or partial response per modified RECIST where a complete response is the disappearance of all target lesions and a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Per RECIST v 1.1, disease progression is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: Time from objective response to 24 months
Population: Because no subjects in Part 2, and only one subject in Part 1, had an objective response the analysis of duration of response was not calculated.
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All serious adverse events that occurred after the subject signed the informed consent form through to the Day 30 Safety Follow-up Visit or 30 days after the last dose of protocol-specified therapy, whichever was later, up to 25 months. All non-serious adverse events that occurred after enrollment through to the Day 30 Safety Follow-up Visit or 30 days after the last dose of protocol-specified therapy, whichever was later, up to 25 months.
Description: Mortality was measured on all subjects. Adverse events were measured on the safety populations (All subjects who received at least one dose of study drug)
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 2 | Part 1 Cohort 3 | Part 2 Cohort 1 | Part 2 Cohort 2 | Part 2 Cohort 3 | Part 2 Cohort 4 | Part 2 Cohort 5 | Part 2 Cohort 6
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 3/3 | 8/15 | 5/8 | 7/16 | 9/16 | 4/9 | 7/16
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 2/3 | 3/15 | 6/7 | 2/16 | 3/16 | 3/9 | 2/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 15/15 | 7/7 | 15/16 | 14/16 | 9/9 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1 (N=3) | Part 1 Cohort 2 (N=3) | Part 1 Cohort 3 (N=3) | Part 2 Cohort 1 (N=15) | Part 2 Cohort 2 (N=7) | Part 2 Cohort 3 (N=16) | Part 2 Cohort 4 (N=16) | Part 2 Cohort 5 (N=9) | Part 2 Cohort 6 (N=15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases To Small Intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Amylase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Bilirubin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1 (N=3) | Part 1 Cohort 2 (N=3) | Part 1 Cohort 3 (N=3) | Part 2 Cohort 1 (N=15) | Part 2 Cohort 2 (N=7) | Part 2 Cohort 3 (N=16) | Part 2 Cohort 4 (N=16) | Part 2 Cohort 5 (N=9) | Part 2 Cohort 6 (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 1 | 0 | 5 | 5 | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adverse Drug Reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 5 | 3 | 1 | 1
Fatigue (General disorders) | 2 | 1 | 1 | 7 | 2 | 1 | 9 | 6 | 3
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Abnormal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 7 | 2 | 2 | 7 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Metastases To Small Intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 2 | 3 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Swelling Face (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 2
Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1
Chills (General disorders) | 0 | 0 | 0 | 6 | 1 | 7 | 4 | 2 | 3
Early Satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Mucous Membrane Disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 4
Vessel Puncture Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Aspartate Aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Amylase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Amylase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood Bilirubin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath Sounds Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Electrocardiogram Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosylated Haemoglobin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematocrit Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Red Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight Fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Eating Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-05-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT00819169/Prot_SAP_000.pdf